CLINICAL TRIAL: NCT06655441
Title: The Effects of 3% Trehalose Ophthalmic Solution on Corneal Epithelial Barrier Function
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Southern California College of Optometry at Marshall B. Ketchum University (Other)
Responsible Party: Principal Investigator, Shora Ansari, Principal Investigator, Southern California College of Optometry at Marshall B. Ketchum University
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: SCCO-Trehalose
Record Dates: First submitted 2024-10-16; First posted 2024-10-23 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Dry Eye Disease (DED)
Keywords: dry eye; trehalose; artificial tears
MeSH Terms: conditions — Dry Eye Syndromes | interventions — Trehalose

STUDY DESIGN:
Intervention Model Description: randomized contralateral eye-controlled trial
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- OS eye receives 3% trehalose drops and OD eye receives control drops (Experimental)
  Interventions: Drug: 3% trehalose
- OD eyes receives 3% trehalose drops and OS eye receives control drops (Other)
  Interventions: Drug: 3% trehalose

INTERVENTIONS:
Drug: 3% trehalose — ophthalmic solution with 3% trehalose in sterile saline in multi dose preservative free bottles

SUMMARY:
The purpose of this research study is to evaluate the effects of trehalose, an ingredient found in commercially available artificial tears, on the corneal barrier function. The investigators will assess corneal dryness and measure the relative corneal epithelial "barrier" function (the degree to which the cornea can prevent penetration of sodium fluorescein dye into the eye) after using eye drops that contain 3% trehalose for one month.

DETAILED DESCRIPTION:
The aim of this study is to recruit moderate to severe dry eye subjects, enroll them in a randomized contralateral eye-controlled trial with an ophthalmic solution containing trehalose 3% in sterile borate buffered saline in one eye and sterile buffered saline in the contralateral eye. The investigators will accomplish this by enrolling a clinic-based sample, undertaking a standardized examination involving signs and symptoms of dry eye, fluorometry, as well as clinical tear and ocular surface measures at baseline and at one-month post-treatment.

ELIGIBILITY:
Inclusion Criteria:

* Adult subjects, > age 18 years, with moderate-to-severe dry eye, defined as fitting criteria for dry eye stages 3 or 4 of the MGD Workshop Management and Treatment subcommittee report.
* Subjects must have normal eyelid position and closure.
* For enrollment as aqueous tear deficiency, subjects must have a Schirmer I result of < 5.0 mm wetting in 5 minutes without anesthesia.

Exclusion Criteria:

* History or evidence of ocular or intraocular surgery in either eye within the past twelve months. LASIK and other kerato-refractive procedure patients can qualify if the most recent surgery or enhancement was 12 or more months prior.
* History or evidence of serious ocular trauma in either eye within the past six months.
* History of hypersensitivity to any component of the study medications.
* History or evidence of epithelial herpes simplex keratitis (dendritic keratitis); vaccinia, active or recent varicella, viral disease of the cornea and/or conjunctiva; chronic bacterial disease of the cornea and/or conjunctiva; mycobacterial infection of the eye; and/or fungal disease of the eye.
* History or evidence of active ocular allergy.
* Females who are pregnant, nursing, or planning a pregnancy during the study.
* Evidence of greater than mild eyelid deformity (e.g., ectropion, entropion, ptosis).
* Use of concomitant topical ocular medications during the study duration.
* Individuals using systemic steroids, immunosuppressive agents and/or anti-cholinergic (e.g. cold and allergy medications, tricyclic antidepressants) for treatment of autoimmune connective tissue disease may not be enrolled in the study if they have not been on a stable dosing regimen for a minimum of 30 days prior to the visit.
* Individuals with uncontrolled diabetes or history or evidence of peripheral neuropathy.
* Active intraocular inflammatory conditions such as iritis.
* Individuals wearing rigid gas permeable or scleral contact lenses within the previous six months of enrollment. Subjects can have worn soft lenses, but not within one month prior to enrollment.
* Individuals using punctual plugs inserted within 30 days of study start.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
corneal epithelial permeability | from enrollment to end of treatment at 4 weeks
  The investigators will measure the relative corneal epithelial barrier function (the degree to which the cornea can prevent penetration of sodium fluorescein dye into the eye) after using eye drops that contain 3% trehalose for one month.

CONTACTS AND LOCATIONS:
Locations (1):
- Marshall B. Ketchum University, Fullerton, California, United States

IPD SHARING:
Plan to Share IPD: Yes
only IPD used in the results publication